CLINICAL TRIAL: NCT02399995
Title: Health Related Quality of Life Following Hepatectomy for Colorectal Liver Metastasis: Global and Disease Specific Changes Over Time
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-057
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Liver Metastasis
Keywords: Quality of Life; Hepatectomy; 15-057

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients following hepatectomy
  Interventions: Behavioral: HRQoL questionnaires.

INTERVENTIONS:
Behavioral: HRQoL questionnaires. — Questionnaires/Forms to be completed preoperatively in clinic with assistance from research study administrator:
  * Baseline sociodemographic and clinical variable data sheet (RSA)
  * EORTC QLQ-C30, QLQ-LMC21, EuroQoL EQ-5D-5L/VAS
  * Baseline disease status and treatment assessment questionnaire Questionnaires/Forms to be completed at first postoperative clinic visit:
  * EORTC QLQ-C30, QLQ-LMC21, EuroQoL EQ-5D-5L/VAS
  Questionnaires/Forms to be mailed to patients at ± 2 month window at the following time points 6,12,18,24, and 36 months following hepatectomy:
  * EORTC QLQ-C30, QLQ-LMC21, EuroQoL EQ-5D-5L/VAS
  * Post surgical follow up disease status and treatment assessment questionnaire
  * At 8 weeks following the mailing of the initial questionnaire package if no response has been received, research personnel will attempt to contact participants by phone.

SUMMARY:
This study is being done to learn more about health related quality of life factors in people having surgery for colorectal liver metastasis. The investigators will look at how these factors may change over time. The information gained from this study will help the investigators to understand the long-term effects that cancer treatments have on the health related quality of life of patients. This information is of high value and will help doctors talk to patients about the possible effects of their operations. While many patients live a long time after such operations, the studies that have been done do not tell the full story of what patients go through after surgery. This study will help us to understand cancer treatment from the patient's perspective. It will also help cancer patients make better decisions about their treatment options and will help them know what to expect after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Colorectal cancer liver metastases (CRLM)
* > 18 years of age
* Absence of unresectable extrahepatic disease
* No previous liver surgery for CRLM
* Clinical risk score (CRS) >/= 3 or > 4 tumors
* CRS includes the following variables;
* Lymph node positive primary
* Disease free interval <12 months
* CEA level >200ng/mL (highest CEA level within 6 months prior to surgery, not including day of surgery)
* Tumor size > 5cm
* Number of tumors >1(based on most recent scan or pathology before liver resection)
* Each variable is given a score of one and summed to give final CRS
* Clinical risk score (CRS) < 3 with pending variables that cannot be determined preoperatively
* If CRS is still < 3 postoperatively, these patients will be excluded and replaced (inevaluable).
* Ability to read and write in English
* Undergoing liver resection/ ablation for CRLM
* Underwent liver resection/ ablation for CRLM, but not their primary tumors

Exclusion Criteria:

* Non-English speaking
* Inability to read and/or write
* International Patients
* Concurrent malignancy (excluding non-melanoma skin cancers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled to undergo liver resection who meet the established criteria will be approached for participation in this study during their preoperative visit. Should patients not undergo their liver resection surgery within 30 days of consent they will be excluded and replaced. Patients undergoing a two stage resection will have their time point frozen for up to six months after their initial surgery. If the time before the second stage of their resection exceeds six months, these patients will be excluded and replaced. The time point will restart at the completion of the second time point. If the patient has an incomplete resection without mention of a second stage resection, the patient will be made ineligible, taken off study, and replaced.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
changes in the quality of life (QoL) | 3 years
  in patients at high risk of recurrence undergoing hepatectomy to assess health related quality of life (HRQoL) using the EORTC QLQ-C30, QLQ-LMC21 and the EuroQol EQ-5D-5L, in patients at high risk of recurrence undergoing hepatectomy for colorectal liver metastasis and to evaluate global and disease specific changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D'Angelica, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and Follow up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow up), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow up), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow up), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Follow Up), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent and follow up), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/